CLINICAL TRIAL: NCT06392204
Title: Assessment of Mandibular CAD/CAM Angle Fracture Reduction/Plate Guide and Customized 3D Grid Plate Versus Champy's Technique (A Randomized Controlled Trial)
Brief Title: CAD/CAM Angle Fracture Reduction/Plate Guide and Customized 3D Grid Plate Versus Champy's Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Arwa Louay Ali Hosni, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSIs
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom made reduction guides and 3D grid plates (Experimental): Mandibular angle fracture reduction and fixation using digitally designed and fabricated patient specific fracture reduction/plate positioning guide and customized 3D grid plate
  Interventions: Procedure: CAD/CAM patient specfifc fracture reduction/plate guide and customized 3D grid plate
- Stock titanium plates (Active Comparator): Mandibular angle fracture reduction and fixation using a single superior border 2.0 miniplate
  Interventions: Procedure: Champy's techqniue

INTERVENTIONS:
Procedure: CAD/CAM patient specfifc fracture reduction/plate guide and customized 3D grid plate — Mandibular angle fracture reduction and fixation using digitally designed and fabricated patient specific fracture reduction/plate positioning guide and customized 3D grid plate
  Arms: Custom made reduction guides and 3D grid plates
Procedure: Champy's techqniue — Mandibular angle fracture reduction and fixation using a single superior border 2.0 miniplate
  Arms: Stock titanium plates

SUMMARY:
This proposed study aims at creating a computer designed patient specific device and titanium plates, that are 3D manufactured in accordance to a preoperative computer aided virtual surgical procedure, aiming to obtain proper alignment of fractured segments of the lower jaw and restore proper teeth positioning therefore overcoming the possible complications of the conventional methods.

Recruited participants will be randomly allocated to a treatment groupp, whether the novel method group or a standard treatment group.

Preoperative panoramic radiograph and a Computed tomography scan will be obtained for each patient.

Surgical procedure will be conducted unde general anesthetic. Medications will be prescribed after surgery and instructions will be given to each patient.

Follow up will be on a weekly basis for the first 6 weeks followed by a followup visit once a month for 6 months.

Postoperative panoramic radiograph and a Computed tomography scan will be obtained at 1 week after the surgical procrdure and again 6 months later.

Digital data obtained from computed tomography scans along with clinical data will be analysed and studied to determine the accuracy of the computer aided device and for comparison with the standard method of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral mandibular angle fracture with or without associated mandibular fractures in need of open reduction and internal fixation.
2. Patients above 18 years old
3. Sufficient dentition to reproduce the occlusal relationships
4. Patient's consent to participate

Exclusion Criteria:

1. Patients with comminuted mandibular angle fracture(s)
2. Patients with any systemic disease that may affect normal healing
3. Patients undergoing chemotherapy or radiotherapy related to the head and neck region
4. Intra-bony lesions in the fracture area that may interfere with proper anatomical reduction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Guide accuracy in repositioning of the fractured segments and in comparison to the preoperative 3D virtual surgical plan. | Outcome will be assessed with preoperative CT (T1-Week 1)immediate postoperative CT at (T3-Week 3)
  Accuracy of postoperative reduction by superimposition of 3D CT data on a 3D specialized software

SECONDARY OUTCOMES:
Postoperative occlusion | Outcome will be assessed clinically at T2 (Week 2) and T3 (Week 3)
  Assessment of postoperative occlusion clinically using a millimeter caliper, occlusion will be categorized into; satisfactory (no gap), mild derangement (gap of 1-2 mm) and deranged (gap more than 2 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt